CLINICAL TRIAL: NCT00779233
Title: A Study to Compare the Relative Bioavailability of Ranbaxy and GlaxoSmithKline Formulation of Zidovudine Tablets 300 mg in Healthy Adult Volunteers Under Fasting Conditions.
Brief Title: Bioequivalence Study of Zidovudine 300 mg Tablets, USP Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 10440303
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence
MeSH Terms: interventions — Zidovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Zidovudine tablets 300 mg of Ranbaxy
  Interventions: Drug: Zidovudine tablets 300 mg
- 2 (Active Comparator): RETROVIR ® 300 mg tablets (GlaxoSmithKline)
  Interventions: Drug: Zidovudine tablets 300 mg

INTERVENTIONS:
Drug: Zidovudine tablets 300 mg

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability of the test formulation of Zidovudine 300 mg tablets with an already marketed reference formulation RETROVIR ® 300 mg tablets (GlaxoSmithKline), under fasted conditions in healthy male and female adult subjects.

DETAILED DESCRIPTION:
A randomized, single dose, two way crossover study was conducted with up to 32 healthy, male and female adult subjects to compare two Zidovudine 300 mg tablet formulations under fasting conditions.

In each period one x 300 mg tablet was administered to fasting subjects. Subjects received the test product in one study period and the reference product in the other period. The order of the treatment administration was as per the dosing randomization schedule. Each dose was separated by at least a 7 day interval.

A total of thirty two (32) subjects (23 males and 9 females) were enrolled for the study, of which only twenty eight (28) subjects completed the clinical portion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18 to 65 years of age, inclusive with a body mass index (BMI) in the range 18-30 kg/m2 inclusive, measured according to Novum Standard operating Procedures
2. Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable method of contraception (e.g. condom with spermicide, IUD, hormonal contraceptives) for at least 30 days prior to dosing and during the duration of the study
3. Good health as determined by lack of clinically significant abnormalities in health assessments performed at screening
4. Signed and dated informed consent form, which meets all criteria of current FDA regulations

Exclusion Criteria:

1. If female, pregnant, lactating or likely to become pregnant during the study
2. History of allergy or sensitivity to Zidovudine, or other antiviral or history of any drug hypersensitivity or intolerance which, in the opinion of the investigator, would compromise the safety of the subject or the study
3. Significant history or current evidence of chronic infectious disease, system disorder or organ dysfunction
4. Presence of gastrointestinal disease or history of malabsorption within the last year
5. History of psychiatric disorders occurring within the last two years that required hospitalization or medication
6. Presence of a medical condition requiring regular treatment with prescription drugs (other than contraceptives)
7. Use of pharmacologic agents known to significantly induce or inhibit drug metabolizing enzymes within 30 days prior to dosing
8. Receipt of any drug as part of research study within 30 days prior to dosing.
9. Drug or alcohol addiction requiring treatment in the past 12 months
10. Donation or significant loss of whole blood (480 mL or more) within 30 days or plasma within 14 days prior to dosing
11. Positive test results for HIV, Hepatitis B surface antigen or Hepatitis C antibody
12. Positive test results for HIV, Hepatitis B surface antigen or Hepatitis C antibody
13. Positive test results for drugs of abuse at screening
14. Positive serum pregnancy test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-09; Primary Completion 2004-09 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Novum Pharmaceutical Research Services, Las Vegas, Nevada, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html